CLINICAL TRIAL: NCT03536299
Title: Measurement and Training of Dual-Task of Gait in Persons With Multiple Sclerosis
Acronym: MS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Texas Woman's University (Other)
Collaborators: TIRR Memorial Hermann (Other); The University of Texas Health Science Center, Houston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20068
Record Dates: First submitted 2018-05-02; First posted 2018-05-24 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Multiple Sclerosis; Gait Disorders, Neurologic; Cognitive Impairment
Keywords: Physical therapy; Gait training; Cognitive-motor interference; Rehabilitation
MeSH Terms: conditions — Multiple Sclerosis; Gait Disorders, Neurologic; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single-Task Gait (Active Comparator): The Single-Task Gait group will be provided with gait training without the Dual-Task cognitive tasks.
  Interventions: Other: Single-task gait
- Dual-Task Gait (Experimental): The Dual-Task Gait group will be provided with gait training AND secondary cognitive tasks during gait training.
  Interventions: Other: Dual-task gait

INTERVENTIONS:
Other: Dual-task gait — During the training sessions, you will participate in gait training with a physical therapist (PT). You will be asked to walk in 2-minute bouts and you will be provided with adequate rest breaks to help manage your fatigue levels. In addition to performing the gait training activities, you will be asked to perform thinking tasks at the same time. These pre-recorded questions or prompts will be provided to you through headphones and a portable music player. This is to help ensure that the PT is able to focus on giving you feedback about your walking ability and answers to the thinking tasks, and on your safety. At the end of each session, you will have walked for a total walking time of 20 minutes.
  Arms: Dual-Task Gait
Other: Single-task gait — During the training sessions, you will participate in gait training with a physical therapist (PT). You will be asked to walk in 2-minute bouts and you will be provided with adequate rest breaks to help manage your fatigue levels. At the end of each session, you will have walked for a total walking time of 20 minutes.
  Arms: Single-Task Gait

SUMMARY:
The purpose of this study is to determine the utility of a performance measure for the dual-task of gait and considering people with multiple sclerosis have both cognitive and motor problems, the secondary aim of this study is to determine the effectiveness of a gait-specific dual-tasking intervention for ambulatory individuals with multiple sclerosis.

DETAILED DESCRIPTION:
A total target sample size of 40 adults with MS and 40 adults without MS will be recruited. The 40 adults without MS will undergo the two baseline testing sessions only for the first phase of the study. 20 of those individuals with MS will be randomly selected to undergo the intervention phase of the study.

The research design will include two groups, the intervention and control group. Both groups will undergo a screening process, two baseline testing sessions, and be randomly assigned to one of the two groups. The duration of the study is 6 weeks in length for a total of 18 training sessions. The intervention group participants will undergo gait training with a specific concomitant cognitive task (dual-task) for a total walking time of 20 minutes and with rest breaks the total session time is ~60 minutes with a physical therapist. The control group will undergo gait training, but without the cognitive task. Feedback from the therapist will be provided to each participant concerning gait mechanics and ways to improve gait regardless of group membership.

Outcome measures data will be collected twice at baseline, once at mid-intervention, once at post-intervention, and once at one-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Ability walk independently with or without an assistive device
* Independent and community-dwelling
* No history or presence of other clinically significant musculoskeletal, cardiovascular, respiratory, or neurologic disease.
* Definite diagnosis of MS [Expanded Disability Status Scale (EDSS) ≤6.5]
* Relapse free for the past 30 days and not currently receiving or will receive any rehabilitation services during the study.

Exclusion Criteria:

- Participants experiencing a true relapse or exacerbation of their symptoms (>24 hours duration in the absence infection or fever, or and ambient increase in body temperature) during the study will be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-05-31 (Actual); Primary Completion 2020-05-31 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Walking and Remembering Test | Week 1, Week 2, Week 5, Week 8, Week 12
  Measures dual-task cost of gait and a titrated forward digit span cognitive task, measured as a percentage.

SECONDARY OUTCOMES:
Change in 2-Minute Walk Test | Week 1, Week 2, Week 5, Week 8, Week 12
  Measures total distance walked by an individual within a 2-minute time period. Measures distance in feet and meters.
Change in 12-Item Multiple Sclerosis Walking Scale | Week 1, Week 2, Week 5, Week 8, Week 12
  Measures self-reported and self-perceived walking disability due to MS in the past 2 weeks. The 12-Item Multiple Sclerosis Walking Scale consists of 12 questions. Each question is rated on a Likert scale from 1 (not at all) to 5 (extremely). The items are scored for a minimum score possible of 12 or a maximal score of 60. This summed score is then divided by 60 and the resulting percentage is interpreted. The scale's final percentage score can range from a minimum of 20% (minimal impact of MS on walking, good outcome) to a maximum of 100% (significant impact of MS on walking, poor outcome).
Change in Fatigue Scale for Motor and Cognitive Functions | Week 1, Week 2, Week 5, Week 8, Week 12
  Measures self-reported physical and mental fatigue levels by the patient with MS. The Fatigue Scale for Motor and Cognitive Functions measures both the motor and cognitive domains of fatigue. The scale consists of 20 total items: 10 items related to motor fatigue and 10 items related to cognitive fatigue. Each item is rated on a Likert scale from 1 (does not apply at all) to 5 (applies completely). The scale items can be summed for a total score (ranging from 20 to 100) or subscales can be summed and interpreted with each subscale ranging from a minimum of 10 points to a maximal 50 points. Higher values in the total score or in the subscale scores indicate worse fatigue and poorer quality of life due to fatigue.
Change in Gait Speed | Week 1, Week 2, Week 5, Week 8, Week 12
  Changes in gait speed (m/s) will be measured for a 10-meter distance. This will be measured by the Protokinetics ZenoWalkway.
Change in Gait Cadence | Week 1, Week 2, Week 5, Week 8, Week 12
  Changes in gait cadence (steps/min) will be measured for a 10-meter distance. This will be measured by the Protokinetics ZenoWalkway.
Change in Step Length | Week 1, Week 2, Week 5, Week 8, Week 12
  Changes in step length (cm) will be measured for a 10-meter distance. This will be measured by the Protokinetics ZenoWalkway.

OTHER OUTCOMES:
Changes in Visual Analog Scale for Fatigue | Week 1, Week 2, Week 5, Week 8, Week 12
  The visual analog scale for fatigue measures immediate self-reported fatigue. This scale is commonly used to monitor and individual's fatigue level to ensure his or her safety during an activity. The individual marks his or her fatigue level on a 10-cm line with one end denoting "no fatigue" and the opposite end denoting "very severe fatigue". The individual's fatigue level is them measured in cm.
Changes in Borg Rating of Perceived Exertion | Week 1, Week 2, Week 5, Week 8, Week 12
  The Borg Rating of Perceived Exertion is a self-reported scale that measures how much exertion an individual is putting forth during a physical activity. It ranges from 6 (no exertion) to 20 (maximal exertion). The individual chooses a number between 6 and 20 to represent his or her level of exertion. This is commonly used to monitor an individual to ensure that he or she is exercising or performing within a safe level.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Brusola, PT,DPT,MSCS, Principal Investigator — Texas Woman's University & TIRR Memorial Hermann
Locations (2):
- United States (2):
  - Texas Woman's University Institute of Health Sciences - Houston Center, Houston, Texas
  - TIRR Memorial Hermann Adult and Pediatric Outpatient Rehabilitation at the Kirby Glen Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No